CLINICAL TRIAL: NCT00301223
Title: An 8-Week Multi-Center, Randomized, Double Blind, Placebo-Controlled Study To Evaluate The Efficacy, Safety And Tolerability Of Pregabalin (150mg-600mg/Day) Using A Flexible Dosing Schedule In The Treatment Of Subjects With Symptoms Of Neuropathic Pain
Brief Title: A Study to Assess the Efficacy, Safety and Tolerability of Pregabalin in Patients With Symptoms of Neuropathic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081081
Record Dates: First submitted 2006-03-07; First posted 2006-03-10 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2011-05

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Pregabalin

SUMMARY:
The objective of this study is to evaluate the efficacy, safety and tolerability for pregabalin using a flexible, optimized dose schedule compared to placebo in relieving the symptoms of neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Chinese outpatient of age 18 to 75
* At screening and baseline, a score of greater than 40 mm on the visual log scale of SF-MPQ

Exclusion Criteria:

* Neurologic disorders unrelated to neuropathic pain, which in the opinion of the investigator, might impair the assessment of pain
* Serum creatinine clearance greater than 60 ml/min

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2006-02; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary efficacy parameter is the endpoint mean pain score based on the pain scores from the subject's daily pain diaries.

SECONDARY OUTCOMES:
The secondary efficacy parameters include the weekly mean pain scores from the subject's daily pain diaries
The Short Form McGill Pain Questionnaire
The Sleep interference score (from subject pain diary)
The Clinician and Patient Global Impression of Change (CGIC and PGIC)
The responder rate defined as the proportion of subjects reporting a decrease of at least 30% in the weekly mean pain scores in each treatment group.
Addtionally, the safety and tolerability of Pregabalin will also be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- China (7):
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Cheng Du Si Chaun
  - Pfizer Investigational Site, Guangzhou
  - Pfizer Investigational Site, Nan Jing, Jiang Su
  - Pfizer Investigational Site, Qing Dao Shan Dong
  - Pfizer Investigational Site, Shanghai
  - Pfizer Investigational Site, Tianjin

REFERENCES:
- [Derived] Schug SA, Parsons B, Almas M, Whalen E. Effect of Concomitant Pain Medications on Response to Pregabalin in Patients with Postherpetic Neuralgia or Spinal Cord Injury-Related Neuropathic Pain. Pain Physician. 2017 Jan-Feb;20(1):E53-E63. PMID 28072797
- [Derived] Markman JD, Jensen TS, Semel D, Li C, Parsons B, Behar R, Sadosky AB. Effects of Pregabalin in Patients with Neuropathic Pain Previously Treated with Gabapentin: A Pooled Analysis of Parallel-Group, Randomized, Placebo-controlled Clinical Trials. Pain Pract. 2017 Jul;17(6):718-728. doi: 10.1111/papr.12516. Epub 2016 Dec 1. PMID 27611736
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081081&StudyName=A+Study+to+Assess+the+Efficacy%2C+Safety+and+Tolerability+of+Pregabalin+in+Patients+with+Symptoms+of+Neuropathic+Pain